CLINICAL TRIAL: NCT00798785
Title: Long-term Function of Beta Cell Allografts in Non-uremic Type 1 Diabetic Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AZ-VUB (Other)
Responsible Party: Principal Investigator, Bart Keymeulen, UZ Brussels, AZ-VUB
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BK_TX_06
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: diabetes mellitus type 1; pancreatic beta cell; transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- group I ATG-MMF-TAC (Experimental): Two clinical implants in the liver:
  First implant: ATG-fresenium Maintained immunosuppression: MMF-TAC n=30
  Interventions: Drug: ATG-MMF-TAC
- group II ATG-Rituximab-MMF-TAC (Experimental): Two clinical implants in the liver:
  First Implant: ATG fresenium + Rituximab Maintained immunosuppression: MMF-TAC n=5
  Interventions: Drug: ATG-Rituximab-MMF-TAC
- group III ATG-Basilixumab-MMF-TAC (Experimental): Two clinical implants in the liver:
  First implant: ATG-fresenium Second implant: basilixumab Maintained immunosuppression: MMF-TAC n=5
  Interventions: Drug: ATG-basilixumab-MMF-TAC
- group IV omentum (Experimental): Two clinical implants: first in the omentum followed by a clinical implant in the liver:
  First implant: ATG-fresenium Maintained immunosuppression: MMF-TAC n=10
  Interventions: Procedure: omentum

INTERVENTIONS:
Drug: ATG-MMF-TAC — ATG-fresenium for max 6 consecutive days depending on CD3 count, starting the day before transplantation.
  Tacrolimus levels for 2 years between 8-10 ng/ml.
  At year 2: randomization:
  group A: till 48 months: tacrolimus levels 8-10 ng/ml 48-60 months: tacrolimus levels 6-8 ng/ml group B: 24-36 months: 6-8 ng/ml 36-60 months: 4-6 ng/ml A subgroup of these patients will receive a sub clinical implant subcutaneous (total n=5) at the time of the first clinical implant in the liver.
  Arms: group I ATG-MMF-TAC
Drug: ATG-Rituximab-MMF-TAC — ATG-fresenium for max 6 consecutive days depending on CD3 count, starting the day before transplantation.
  Rituximab: the day before transplantation, day 5; 12 and 19 after implantation. Tacrolimus levels for 2 years between 8-10 ng/ml.
  At year 2: randomization:
  group A: till 48 months: tacrolimus levels 8-10 ng/ml 48-60 months: tacrolimus levels 6-8 ng/ml group B: 24-36 months: 6-8 ng/ml 36-60 months: 4-6 ng/ml A subgroup of these patients will receive a sub clinical implant, subcutaneous at the time of the first clinical implant in the liver.
  Arms: group II ATG-Rituximab-MMF-TAC
Drug: ATG-basilixumab-MMF-TAC — First transplantation:
  ATG-fresenium for max 6 consecutive days depending on CD3 count, starting the day before transplantation.
  Second transplantation:
  Basilixumab:
  the day before the second transplantation followed by 4days after transplantation.
  Tacrolimus levels for 2 years between 8-10 ng/ml.
  At year 2: randomization:
  group A: till 48 months: tacrolimus levels 8-10 ng/ml 48-60 months: tacrolimus levels 6-8 ng/ml group B: 24-36 months: 6-8 ng/ml 36-60 months: 4-6 ng/ml A subgroup of these patients will receive a sub clinical implant, subcutaneous at the time of the first clinical implant in the liver.
  Arms: group III ATG-Basilixumab-MMF-TAC
Procedure: omentum — Two clinical implants: first in omentum followed by a clinical implant in the liver:
  In a group of 10 patients, a clinical implant in the omentum will be implanted. If random C-peptide levels >= 0.5 ng/ml are measured at 2 months post-transplantation, a second omental implant will be done. If no clinical relevant beta cell graft function is measured, two intraportal implants will be given as a compassionate use procedure. An interim analysis after 5 patients has to shown clinical relevant function at month 2 in 3 out of 5 patients before the subsequent 5 patients can be transplanted in the omentum.
  Arms: group IV omentum

SUMMARY:
The present proof of concept study addresses the following specific aims:

The general objectives of this work are:

1. To increase and maintain the functional beta-cell mass after islet transplantation under a condition of low-dose tacrolimus
2. To co-investigate the potential of alternative sites for encapsulated beta-cells

DETAILED DESCRIPTION:
1. Aim 1: To increase functional beta cell mass by adding rituximab at first implantation
2. Aim 2: To increase functional beta cell mass by adding basilixumab at second implantation
3. Aim 3: To assess the influence of down-tapering the tacrolimus dose during posttransplant years 2-5 on these data, on metabolic control, on the prevalence of hypoglycemia and on safety parameters.
4. Aim 4: To investigate the potential of the peritoneum and omentum as an alternative site for encapsulated beta-cells.
5. Aim 5: To investigate the potential of the brachioradial muscle as an alternative site for encapsulated beta-cells.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years, male or female, Caucasian or not; only subjects < 50 yrs will be allocated to the rituximab treatment arm
* Body weight < 100 kg; patients with a bodyweight of < 80kg, will receive priority
* Patients with a BMI ≤ 27 kg/m2 will receive priority
* Type 1 insulin-dependent diabetes
* C-peptide < 0.07 nmol/l (<0.2 µg/l) 6 min. after glucagon IV (1mg) (glycemia > 180 mg/dl)
* Intensive insulin therapy for more than two years, patients with insulin pump during at least 2 months before inclusion will receive priority
* Patients should have at least one of the following chronic complications of diabetes:

  * Plasma creatinine <2 mg/dl and albuminuria 30-1000 mg/ 24hrs on 3 separate determinations (>1 month) outside an episode of illness, despite intake of ACE inhibitors; mean systolic blood pressure should be under 130 mmHg and mean diastolic blood pressure under 85 mmHg, when measured at home with ambulatory BP monitoring
  * Moderate or severe non-proliferative or proliferative retinopathy
  * Hypoglycemic unawareness
* Cooperative and reliable patient giving informed consent by signature

Exclusion Criteria:

* Smoker
* EBV antibody negativity
* HIV 1 & 2 antibody positivity
* CMV IgM positivity
* Plasma creatinine ≥ 2 mg/dl and/or albuminuria ≥1000 mg/24 hrs
* History of thrombosis or pulmonary embolism
* History of malignancy, tuberculosis or chronic viral hepatitis
* History of any other serious illness which could be relevant for the protocol
* Presence of HLA antibodies
* Blood donation within one month prior to screening or during the study
* Symptoms and/or signs of infection, particularly (present or past) endocarditis, osteomyelitis, past tuberculosis with requirement for therapy
* Any history of hepatic or neoplastic disease
* Any history of renal disease (except diabetes)
* Abnormal liver function tests and /or NMR of liver
* Hemoglobinopathy
* History of any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risks to the patient
* Pregnancy or use of inadequate contraception by female patients of childbearing potential
* Use of illicit drugs or overconsumption of alcohol (> 3 beers/day) or history of drug or alcohol abuse
* Being legally incapacitated, having significant emotional problems at the time of the study, or having a history of psychiatric disorders
* Having received antidepressant medications during the last 6 months
* Having participated the last 12 months or participating in another clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-10; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Evidence of clinically relevant beta cell graft function | up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Bart Keymeulen, MD PhD, Principal Investigator — University Hospital Brussel
Locations (4):
- Belgium (4):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - University Hospital Brussels, Brussels
  - Hopital Erasme, Brussels
  - University Hospital Leuven, Leuven

REFERENCES:
- [Background] Keymeulen B, Gillard P, Mathieu C, Movahedi B, Maleux G, Delvaux G, Ysebaert D, Roep B, Vandemeulebroucke E, Marichal M, In 't Veld P, Bogdani M, Hendrieckx C, Gorus F, Ling Z, van Rood J, Pipeleers D. Correlation between beta cell mass and glycemic control in type 1 diabetic recipients of islet cell graft. Proc Natl Acad Sci U S A. 2006 Nov 14;103(46):17444-9. doi: 10.1073/pnas.0608141103. Epub 2006 Nov 7. PMID 17090674
- [Background] Movahedi B, Keymeulen B, Lauwers MH, Goes E, Cools N, Delvaux G. Laparoscopic approach for human islet transplantation into a defined liver segment in type-1 diabetic patients. Transpl Int. 2003 Mar;16(3):186-90. doi: 10.1007/s00147-002-0517-7. Epub 2003 Feb 15. PMID 12664214
- [Background] Maleux G, Gillard P, Keymeulen B, Pipeleers D, Ling Z, Heye S, Thijs M, Mathieu C, Marchal G. Feasibility, safety, and efficacy of percutaneous transhepatic injection of beta-cell grafts. J Vasc Interv Radiol. 2005 Dec;16(12):1693-7. doi: 10.1097/01.RVI.0000182506.88739.39. PMID 16371537
- [Derived] Lee D, Gillard P, Hilbrands R, Ling Z, Van de Velde U, Jacobs-Tulleneers-Thevissen D, Maleux G, Lapauw B, Crenier L, De Block C, Mathieu C, Pipeleers D, Keymeulen B. Use of Culture to Reach Metabolically Adequate Beta-cell Dose by Combining Donor Islet Cell Isolates for Transplantation in Type 1 Diabetes Patients. Transplantation. 2020 Oct;104(10):e295-e302. doi: 10.1097/TP.0000000000003321. PMID 32433237
- [Derived] Balke EM, Demeester S, Lee D, Gillard P, Hilbrands R, Van de Velde U, Van der Auwera BJ, Ling Z, Roep BO, Pipeleers DG, Keymeulen B, Gorus FK. SLC30A8 polymorphism and BMI complement HLA-A*24 as risk factors for poor graft function in islet allograft recipients. Diabetologia. 2018 Jul;61(7):1623-1632. doi: 10.1007/s00125-018-4609-z. Epub 2018 Apr 20. PMID 29679103
- [Derived] Lee D, Keymeulen B, Hilbrands R, Ling Z, Van de Velde U, Jacobs-Tulleneers-Thevissen D, Maleux G, Lapauw B, Crenier L, De Block C, Mathieu C, Pipeleers D, Gillard P. Age and Early Graft Function Relate With Risk-Benefit Ratio of Allogenic Islet Transplantation Under Antithymocyte Globulin-Mycophenolate Mofetil-Tacrolimus Immune Suppression. Transplantation. 2017 Sep;101(9):2218-2227. doi: 10.1097/TP.0000000000001543. PMID 27779572